CLINICAL TRIAL: NCT06168084
Title: Rescue Therapy for Helicobacter Pylori Eradication: A Randomized and Non-inferiority Trail of Vonorazon and Amoxicillin Dual Therapy Versus Bismuth-containing Quadruple Therapy
Brief Title: Helicobacter Rescue Therapy With Vonorazon and Amoxicillin Dual Therapy Versus Bismuth-containing Quadruple Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yongquan Shi (Other)
Responsible Party: Sponsor-Investigator, Yongquan Shi, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20232236-F-2
Record Dates: First submitted 2023-12-04; First posted 2023-12-13 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Gastritis Dyspepsia Helicobacter Pylori Infection Gastric Cancer Peptic Ulcer
MeSH Terms: interventions — 1-(5-(2-fluorophenyl)-1-(pyridin-3-ylsulfonyl)-1H-pyrrol-3-yl)-N-methylmethanamine; Amoxicillin; Bismuth; Esomeprazole; Tetracycline; Furazolidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Vonorazon and amoxicillin dual therapy (Experimental): Vonorazon 20 mg daily for 14 days # amoxicillin 1000 mg by mouth three time daily for 14 days
  Interventions: Drug: Vonoprazan; Drug: amoxicillin
- Bismuth-containing quadruple therapy (Active Comparator): Tetracycline 500mg three time daily for 14 days#furazolidone 100 mg, esomeprazole 40 mg, and Bismuth 220mg by mouth, twice daily for 14 days.
  Interventions: Drug: Bismuth; Drug: Esomeprazole; Drug: Tetracycline; Drug: Furazolidone

INTERVENTIONS:
Drug: Vonoprazan — Vonoprazan and amoxicillin dual therapy:given for 14 days at a dose of vonoprazan 20mg 1 tablet BID plus amoxicillin 500 mg 2 capsules TID
  Arms: Vonorazon and amoxicillin dual therapy
Drug: amoxicillin — Vonoprazan and amoxicillin dual therapy:given for 14 days at a dose of vonoprazan 20mg 1 tablet BID plus amoxicillin 500 mg 2 capsules TID
  Arms: Vonorazon and amoxicillin dual therapy
Drug: Bismuth — Bismuth-containing quadruple therapy: given for 14 days at a dose of bismuth 110 mg 2 capsules BID plus esomeprazole 20 mg 2 tablets BID#tetracycline 250mg 2 capsules TID and furazolidone 100mg 1 tablets BID
  Arms: Bismuth-containing quadruple therapy
Drug: Esomeprazole — Bismuth-containing quadruple therapy: given for 14 days at a dose of esomeprazole 20mg 2 tablets BID plus bismuth 110 mg 2 capsules BID#tetracycline 250mg 2 capsules TID and furazolidone 100mg 1 tablets BID
  Arms: Bismuth-containing quadruple therapy
Drug: Tetracycline — Bismuth-containing quadruple therapy:given for 14 days at a dose of tetracycline 250mg 2 capsules TID plus furazolidone 100mg 1 tablets BID#esomeprazole 20 mg 2 tablets BID and bismuth 110 mg 2 capsules BID
  Arms: Bismuth-containing quadruple therapy
Drug: Furazolidone — Bismuth-containing quadruple therapy:given for 14 days at a dose of furazolidone 100mg 1 tablets BID plus tetracycline 250mg 2 capsules TID#esomeprazole 20 mg 2 tablets BID and bismuth 110 mg 2 capsules BID
  Arms: Bismuth-containing quadruple therapy

SUMMARY:
This study aims at evaluating efficacy and safety of Vonorazon and amoxicillin dual therapy versus bismuth-containing quadruple Therapy(bismuth#esomeprazole#tetracycline and furazolidone) in H. pylori rescue therapy. It is hypothesized that Vonorazon and amoxicillin dual therapy is non-inferior to bismuth-containing quadruple Therapy. Patients with confirmed failure of H. pylori eradication will be randomized to one of the treatments described above. At week 6 follow-up visits, a urea breath test#rapid urease test or helicobacter pylori stool antigen test will be performed to confirm eradication.

DETAILED DESCRIPTION:
The study will include three phases: screening, treatment and follow-up. Screening: this phase will last a maximum of 14 days and subjects eligibility will be evaluated after signing informed consent. One of urea breath test#rapid urease test or helicobacter pylori stool antigen test will be performed in addition to the baseline routine evaluations.

Treatment: Subjects are randomly assigned to treatment and will be treated for 14 days. A randomization visit will take place on Day 0 and an end-of-treatment visit will take place between day 14 and 16.

Follow-up: includes one visits. Approximately 28 days after the end of treatment. Eradication of H. Pylori will be confirmed by one of urea breath test#rapid urease test or helicobacter pylori stool antigen test.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age between 18~70, both gender. 2. Patients who had failed H.pylori eradication therapies . 3. Women are eligible if they are not pregnant or nursing, and if they are of childbearing potential they are required to use medically acceptable contraception for the duration of the study and 30 days thereafter.

Exclusion Criteria:

* 1. Patients who have previously used tetracycline and furazolidone antibiotics to eradicate infection with H. pylori.

  2. Contraindications to study drugs. 3. Substantial organ impairment, severe or unstable cardiopulmonary or endocrine disease.

  4. Constant use of anti-ulcer drugs ( including taking proton-pump.inhibitors(PPI) within 2 weeks before the [13C] urea breath test), antibiotics or bismuth complexes (more than 3 times /1 month before screening).

  5. Pregnant or lactating women. 6. Underwent upper gastrointestinal Surgery. 7. Dysphagia. 8. Evidence of bleeding or iron efficiency anemia. 9. A history of malignancy. 10. Drug or alcohol abuse history in the past 1 year. 11. Systemic use of corticosteroids, non steroidal anti-inflammatory drugs, anticoagulants, platelet aggregation inhibitors (except the use of aspirin for less than 100 mg/d).

  12. Mental disorder. 13. Enrolled in other clinical trials in the past 3 months. 14. Refuse to sign informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Actual)
Dates: Start 2023-06-06 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori eradication | 28 days after treatment
  The primary end point of this study is H.pylori eradication#established by negative [13C] urea breath test #DOB value below 3.9#28 days after the end of eradication

SECONDARY OUTCOMES:
symptoms effective rates | 14 days of treatment, and 28 days after treatment
  symptoms improvement rates Evaluation improvement rate of symptoms 2 weeks of treatment and 4 weeks after the end of treatment. Symptom improvement rate =# t total score before treatment - total score after treatment#/total score before treatment x100%. Total score = frequency + severity.Frequency score is calculated by all the frequency of heartburn, reflux, abdominal pain, and flatulence, etc. Severity is accumulated by the degree of symptoms described above, which is divided to 4 degree as 0 presenting none, and 3 presenting most severe
adverse events | 14 days of treatment, and 28 days after treatment
  Participants with Adverse Events as a Measure of Safety and Tolerability.The common side effects of the study include headache,dizziness,skin rash,other gastrointestinal disorders,pyrexia,cough and back pain.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Xijing Hosipital of Digestive Disease, Xi'an, Shaanxi
  - Xijing Hosipital of Digestive Disease, Xi’an, Shanxi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang J, Wang X, Song S, Zhu X, Lv T, Wang L, Lei L, Wang Y, Lei Y, Wang Y, Zhu X, Zhang L, Chen M, Shi Y. Efficacy and Safety of Vonoprazan and High-Dose Amoxicillin Dual Therapy for Rescue Treatment of Helicobacter pylori Infection: A Multicenter Randomized Controlled Trial. United European Gastroenterol J. 2025 Oct;13(8):1541-1549. doi: 10.1002/ueg2.70070. Epub 2025 Jun 21. PMID 40543051